CLINICAL TRIAL: NCT02885415
Title: Prevalence of Myocardial Injury in Gastrointestinal Surgery Patients - A Multi-center Prospective Cohort Study - POMY
Brief Title: Prevalence of Myocardial Injury in Gastrointestinal Surgery Patients
Acronym: POMY
Status: Completed | Type: Observational
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Midland Regional Hospital, Tullamore (Other); Mayo University Hospital (Unknown); Letterkenny University Hospital (Unknown); University College Hospital Galway (Other)
Responsible Party: Principal Investigator, KHALID AHMED, Mr, National University of Ireland, Galway, Ireland
Other Study IDs: C.A 1518
Record Dates: First submitted 2016-08-08; First posted 2016-08-31 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Myocardial Injury
MeSH Terms: interventions — Digestive System Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Gastrointestinal surgery — Major resectional gastrointestinal surgery (define as resection of part of gastrointestinal tract during esophageal, Gastric or colorectal surgeries)

SUMMARY:
the troponin level and ECGs pre and post operative will be used to determined prevalence of myocardial injury among patients undergoing gastrointestinal surgery

DETAILED DESCRIPTION:
AIM:

The aim of this study is to determine the prevalence of myocardial injury in gastrointestinal surgery patients and to establish baseline data to allow evaluation of the potential benefit of RIPC (remote ischemic preconditioning) in these patients

Significance:

In available literature was one study including 51 patients that focused on postoperative arrhythmias in colorectal surgery . We think this study is important to establish more specifically the prevalence of myocardial injury in this cohort of patients so we can measure in our future research if RIPC or any other protective method could produce significant effect.

Study Design:

Prospective Observational cohort Study

Study Objectives:

To determine the prevalence of myocardial injury in patients undergoing gastrointestinal surgery

Patients and Locations:

Patients older than 18 years undergoing major resectional gastrointestinal surgery in Galway University Hospitals (UCHG, Mayo university Hospital), The Midland Regional Hospital, Tullamore and Letterkenny University Hospital will be asked to join the study and will considered eligible after informed consent and information handouts provided.

Protocol:

After informed consent patients' pre-op demographic data, co-morbidities, bloods including troponin and ECG will be recorded. Serum troponin levels will be measured daily for the first 72 hours and a 12-lead electrocardiogram will be performed at 48 hours post-surgery. There will be 1 year flow up for candidates

Data Handling:

The data for each hospital will be kept locally and patients will be allocated numbers for later data analysis. The pooled data will be analyzed using a secure computer in an NUI Galway research facility building. No patients' name or any other identifier will be associated with this data except for their study number assigned earlier

Primary Outcome:

Prevalence of myocardial injury by comparing pre and post-op troponin and ECGs. The diagnosis of myocardial injury will be determined by a cardiologist after examining troponin and ECGs results using SAVES trial criteria (5).

Perioperative Myocardial injury will include silent myocardial infarctions as determined by the study cardiologist upon examination of study ECGs and troponin results. The diagnosis of a myocardial injury will require the presence of at least two of the following:

1. Characteristic ischemic symptoms lasting at least 20 minutes
2. Electrocardiographic changes including acute ST elevation followed by the appearance of Q waves or the loss of R waves, the development of new left bundle branch block, new persistent T wave inversion lasting at least 24 hours or new ST segment depression persisting over 24 hours
3. Positive troponin above normal range (0-14)
4. New-onset arrhythmia (ventricular or supraventricular tachycardia or fibrillation) with an associated rise in troponin levels
5. Alternatively, myocardial injury will be recorded if the patient develops sudden unexpected cardiac death involving cardiac arrest with symptoms suggestive of myocardial ischemia and accompanied by presumably new ST elevation or new left bundle branch block and/or fresh thrombus on coronary angiography and/or at post-mortem, but death occurring before blood samples could be obtained or at a time before the appearance of cardiac troponin I or T in the blood.

Other Data:

* Age
* Gender
* Procedure type
* Renal Profile (Renal impairment will be consider when interpreting Troponin values)
* ECG
* Ethnicity
* Diabetes
* BP
* History of Cardiac event
* Other Comorbidities
* Smoking history
* NYHA classification (New York Heart Association )
* Medication at time of consent (Blood pressure and heart rate control medications)

Exclusion Criteria

* Documented Pre-op Myocardium Injury
* Refused or unable to give informed consent
* Laparoscopic fundoplication
* Laparoscopic cholecystectomy surgery
* Appendectomy surgery
* Hernia repair surgery

Sample Size:

This is a prospective study to determine the incidence of myocardial injury in gastrointestinal surgical patients. There are no existing data upon which to base a sample size calculation. We estimate that data from 100 patients should provide a sufficient sample size to generate a reasonably robust incidence estimate. However, if the included centers recruit more patients they will be included in our analysis

Statistical Analysis:

Statsdirect will be used for analysis of the study results Budget No additional budget for the study will be needed as tests required routinely requested within the study clinical setting. The analysis and management of the study will be performed by clinical research fellow funded by National University of Ireland Galway

Conflict of interest:

Study team declare no conflict of interest

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years undergoing major resectional gastrointestinal surgery (define as resection of part of gastrointestinal tract ( oesophageal, Gastric or colorectal surgeries)

Exclusion Criteria:

* - Documented Pre-op Myocardium Injury
* Refused or unable to give informed consent
* Laparoscopic fundoplication
* Laparoscopic cholecystectomy surgery
* Appendectomy surgery
* Hernia repair surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years undergoing major resectional gastrointestinal surgery in Galway University Hospitals (UCHG, Mayo university Hospital), The Midland Regional Hospital, Tullamore and Letterkenny University Hospital will be asked to join the study and will considered eligible after informed consent and information handouts provided.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08-05 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Change in Troponin | Pre-Op and 3 days series post-op results
  Cahnges in Troponin levels Pre-Op and Day 1, Day 2 and Day 3 post-OP
ECG changes | Pre-Op and 48 hours post-op
  Changes as per Protocol Criteria

CONTACTS AND LOCATIONS:
Locations (4):
- Ireland (4):
  - University Collage Hospital Galway, Galway, Co Galway
  - Letterkenny University Hospital, Letterkenny, Donegal
  - Mayo University Hospital, Castlebar, Mayo
  - Midland Regional Hospital, Tullamore, Tullamore

IPD SHARING:
Plan to Share IPD: No